CLINICAL TRIAL: NCT03777579
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled Study of JS001 (Anti-PD-1 Antibody) in Combination With Nab-Paclitaxel Compared With Placebo With Nab-Paclitaxel as First-line Therapy for Patients With Primarily Diagnose or Recurrent and Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of First-line JS001 and Nab-paclitaxel Versus Palcelbo and Nab-Paclitaxel in Participants With Advanced Recurrent or Metastatic TNBC
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: trial handovered to another sponser.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NABP201801
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2018-12

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 Plus Nab-Paclitaxel (Experimental): Participants assigned to JS001 plus nab-paclitaxel will receive both agents until disease progression or unacceptable toxicity.
  Interventions: Drug: JS001，an engineered anti-PD-1 antibody; Drug: Nab-Paclitaxel
- Placebo Plus Nab-Paclitaxel (Placebo Comparator): Participants assigned to placebo plus nab-paclitaxel will receive both agents until disease progression or unacceptable toxicity.
  Interventions: Drug: Nab-Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: JS001，an engineered anti-PD-1 antibody — JS001 at a fixed dose of 240 milligrams via intravenous (IV) infusion on Days 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Other Names: Terepril monoclonal antibody
  Arms: JS001 Plus Nab-Paclitaxel
Drug: Nab-Paclitaxel — Nab-Paclitaxel at a starting dose of 125mg per square meter via IV infusion on Days 1, 8 of each 21-day cycle. Nab-Paclitaxel will be administered until disease progression or unacceptable toxicity.
  Other Names: Paclitaxel For Injection（Albumin Bound）
Drug: Placebo — Placebo administered via intravenous (IV) infusion on Days 1 of each 21-day cycle until disease progression or unacceptable toxicity.
  Arms: Placebo Plus Nab-Paclitaxel

SUMMARY:
This multicenter, randomized, double-blind study will evaluate the efficacy, safety of JS001 administered with nab-paclitaxel compared with placebo in combination with nab-paclitaxel as first-line therapy in participants with primarily diagnosed stage IV and recurrent or metastatic triple-negative breast cancer (TNBC) who have not received prior systemic therapy for metastatic breast cancer (mBC).

ELIGIBILITY:
Inclusion Criteria:

1. Primarily diagnosed stage IV or recurrent and metastatic, histologically documented TNBC characterized by absence of human epidermal growth factor 2 (HER2), estrogen receptor (ER), and progesterone receptor (PR) expression;
2. No prior chemotherapy or targeted systemic therapy for inoperable stage IV or metastatic TNBC；
3. Eligible for taxane monotherapy；
4. Eastern Cooperative Oncology Group performance status of 0 or 1；
5. Measurable disease as defined by RECIST v1.1；
6. Adequate hematologic and end-organ function。

Exclusion Criteria:

1. Known central nervous system (CNS) disease with active syndrome or untreated disease, except for treated asymptomatic CNS metastases；
2. History of autoimmune disease；
3. History of Anaphylaxis to PD-(L)1 antibody or CTLA-4 antibody or paclitaxel;
4. Prior allogeneic stem cell or solid organ transplantation;
5. Active hepatitis B or hepatitis C;
6. Positive of HIV antibody.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)by Independent Review Committee (IRC) | From Day 1 to disease progression (PD) or death from any cause, assessed up to end of study (up to approximately 30 months)
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Assessed Using RECIST v1.1 by investigator | From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 30 months)
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Objective response rate (ORR) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)by IRC | From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 30 months)
  ORR is defined as the rate of CR or PR, as determined by IRC using RECIST v1.1 criteria.
Duration of response (DoR) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)by IRC | From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 30 months)
  DoR is defined as the time period from the date of initial CR or PR until the date of PD or death from any cause, whichever occurs first.
Disease control rate (DCR) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)by IRC | From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 30 months)
  DCR is defined as the rate of of CR, PR, or stable disease according to RECIST v1.1.
Overall Survival (OS) | From Day 1 to death from any cause, assessed up to end of study (up to approximately 30 months)
  OS is defined as the time from randomization to death from any cause.
OS rate at 12 months | the percent of participants that are alive at 12months from Day 1.
  OS is defined as the time from randomization to death from any cause.
OS rate at 24 months | the percent of participants that are alive at 24 months from Day 1.
  OS is defined as the time from randomization to death from any cause.
PFS Assessed Using immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) by investigator | From Day 1 to death from any cause, assessed up to end of study (up to approximately 30 months)
  Progression is confirmed in the target lesion category if the next imaging assessment after iUPD (4-8 weeks later) confirms a further increase in sum of measures of target disease from iUPD, with an increase of at least 5mm.
ORR Assessed Using immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) by investigator | From Day 1 to death from any cause, assessed up to end of study (up to approximately 30 months)
  ORR is defined as the rate of iCR or iPR, as determined by investigator using iRECIST criteria.
DoR Assessed Using immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) by investigator | From Day 1 to death from any cause, assessed up to end of study (up to approximately 30 months)
  DoR is defined as the time period from the date of initial iCR or iPR until the date of iCPD or death from any cause, whichever occurs first.
DCR Assessed Using immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) by investigator | From Day 1 to death from any cause, assessed up to end of study (up to approximately 30 months)
  DCR is defined as the rate of of iCR, iPR, or stable disease according to iRECIST.
Percentage and severity of Participants With Adverse Events (AEs) | From Day 1 to 60 days after last dose of study drug, assessed up to end of study (up to approximately 30 months)
  percentage and CTC AE(v5.0) of AEs
Percentage of Participants With Anti-Drug Antibodies (ATAs) | Pre-dose (60minutes±10minutes) on Day 1 of Cycles 1, 3, 5, 7, 9 and at every 6 cycles thereafter until disease progression, at disease progression. (maximum up to 30 months) (1 Cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: JIANG ZE FEI, PHD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The fifth medical center of PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Z, Ouyang Q, Sun T, Zhang Q, Teng Y, Cui J, Wang H, Yin Y, Wang X, Zhou X, Wang Y, Sun G, Wang J, Zhang L, Yang J, Qian J, Yan M, Liu X, Yi T, Cheng Y, Li M, Zang A, Wang S, Wang C, Wu X, Cheng J, Li H, Lin Y, Geng C, Gu K, Xie C, Xiong H, Wu X, Yang J, Li Q, Chen Y, Li F, Zhang A, Zhang Y, Wu Y, Nie J, Liu Q, Wang K, Mo X, Chen L, Pan Y, Fu P, Zhang H, Pang D, Sheng Y, Han Y, Wang H, Cang S, Luo X, Yu W, Deng R, Yang C, Keegan P. Toripalimab plus nab-paclitaxel in metastatic or recurrent triple-negative breast cancer: a randomized phase 3 trial. Nat Med. 2024 Jan;30(1):249-256. doi: 10.1038/s41591-023-02677-x. Epub 2024 Jan 8. PMID 38191615